CLINICAL TRIAL: NCT00140569
Title: Randomized Study for Patients With Follicular Lymphoma Needing Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lymphoma Study Association (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Gelf-94
Record Dates: First submitted 2005-08-31; First posted 2005-09-01 (Estimated); Last update posted 2005-09-01 (Estimated); Status verified 2005-08

CONDITIONS: Follicular Lymphoma
Keywords: follicular lymphoma; CHVP + interferon; fludarabine; autotransplant
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Interferons; fludarabine; Whole-Body Irradiation; Transplantation, Autologous

INTERVENTIONS:
Procedure: CHVP + interferon
Drug: fludarabine
Procedure: CHOP + TBI and autotransplant

SUMMARY:
2 parallel studies.

* For young patients (18-60 years): randomization between CHVP + interferon for 18 months and 4 CHOP followed by autotransplant after TBI
* For elderly patients (>60 years): randomization between CHVP + interferon for 18 months and fludarabine 5 days every months for 6 months

DETAILED DESCRIPTION:
2 parallel studies.

* For young patients (18-60 years): randomization between CHVP + interferon for 18 months and 4 CHOP followed by autotransplant after TBI
* For elderly patients (>60 years): randomization between CHVP + interferon for 18 months and fludarabine 5 days every months for 6 months

ELIGIBILITY:
Inclusion Criteria:

* study 1 (young patients): being less than 61 years old with a follicular lymphoma and needing to be treated because of high LDH level, high beta-2 microglobulin level, poor performance status, or large tumoral mass (lymph node >7 cm, symptomatic splenomegaly, pleura effusion, or sign of compression by the tumor mass)
* study 2 (elderly patients): being older than 60 years with a follicular lymphoma and needing to be treated because of high LDH level, high beta-2 microglobulin level, poor performance status, or large tumoral mass (lymph node >7 cm, symptomatic splenomegaly, pleura effusion, or sign of compression by the tumor mass)

Exclusion Criteria:

* contra-indication to anthracycline or interferon
* transformation into large cell lymphoma
* previous treatment
* localized stage without criteria of large tumor mass
* patients HIV+

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 1994-01; Study Completion 2004-01

PRIMARY OUTCOMES:
Progression-free survival

SECONDARY OUTCOMES:
Overall survival
Toxicity
Response rates

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand Coiffier, MD, Study Chair — Hospices Civils de Lyon; Catherine Sebban, MD, Principal Investigator — Centre Leon Berard
Locations (8):
- Groupe d'atude des lymphome de l'adulte, Yvoir, Belgium
- France (7):
  - Hôpital Henri Mondor, Créteil
  - Centre Léon Bérard, Lyon
  - Hôpital Saint Louis, Paris
  - Service d'Hématologie - Centre Hospitalier Lyon-Sud, Pierre-Bénite
  - Centre Hospitalier Robert Debré, Reims
  - Centre Henri Becquerel, Rouen
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Result] Coiffier B, Neidhardt-Berard EM, Tilly H, Belanger C, Bouabdallah R, Haioun C, Brice P, Peaud PY, Pico JL, Janvier M, Solal-Celigny P, Brousse N. Fludarabine alone compared to CHVP plus interferon in elderly patients with follicular lymphoma and adverse prognostic parameters: a GELA study. Groupe d'Etudes des Lymphomes de l'Adulte. Ann Oncol. 1999 Oct;10(10):1191-7. doi: 10.1023/a:1008347425795. PMID 10586336
- See also: Official site of the Groupe d'Etudes des Lymphomes de l'Adulte (In french) — http://www.gela.org